CLINICAL TRIAL: NCT06105047
Title: Validation of a Remediation Method for Memory Disorders Using Motor and Emotional Encoding in Patients With Alzheimer's Disease (AD)
Brief Title: Validation of a Remediation Method for Memory Disorders Using Motor and Emotional Encoding in Patients With Alzheimer's Disease
Acronym: ADAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23CH154; ANSM (Other: 2023-A01403-42)
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Action memory; Musical memory
MeSH Terms: conditions — Alzheimer Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Alzheimer disease (Experimental): Patients will perform experimental task in four conditions : control, mime, emotion, dual
  Interventions: Behavioral: Cognitive tests

INTERVENTIONS:
Behavioral: Cognitive tests — . Patients will perform experimental task in four conditions : control, mime, emotion, dual In a control condition : they will be asked to read the sentence aloud; in a motor-only condition, they will also be asked to mime the sentence; in an emotional-only condition, they will be asked to read the sentence while listening to music; in a dual condition, they will be asked to both mime and listen to music. Immediately after each condition, they will realize a recognition task
  * quiz : Geneva Music Induced Checklist, GMIAC, Coutinho & Scherer, 2017

SUMMARY:
Memories are more robust when they are multitraced. This means that the more a piece of information is mediated by different sensory inputs, the more resistant it is to being forgotten. Many works in the field of embodied cognition show that new learnings are better recalled over the long term when they are learned during body mobilization. Other works show that musical stimulation could be a good way of eliciting physiological and emotional states more favorable to the memorization of new contents. However, to date, no studies have examined the positive effects of these two tools combined in Alzheimer's disease. The investigators suggest that it is possible to optimize memory in Alzheimer's disease by referring to their motor and emotional resources. The hypothesis is that information will be better recalled with multimodal enriched learning.

DETAILED DESCRIPTION:
In a within subjects design, all patients take part in four conditions. In each condition, sentences describing actions will be displayed. In a control condition, they will be asked to read the sentence aloud; in a motor-only condition, they will also be asked to mime the sentence; in an emotional-only condition, they will be asked to read the sentence while listening to music; and in a dual condition, they will be asked to both mime and listen to music. Immediately after each condition, they will realize a recognition task. The main criterion used in our statistical analyses will be the discrimination threshold.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease by one of the consulting physicians, neurologist and/or geriatrician of whom the patient has been informed.
* Early stage (MMSE ≥ 22)
* Neuropsychological assessment within 6 months of inclusion.
* Affiliation with a social security scheme
* Age equal to or greater than 60
* French mother tongue
* Agreement to participate / signature of consent form

Exclusion Criteria:

* Uncorrected perceptual disorders
* Other neurological or psychiatric history
* Inability to communicate
* Delusional or psychotic state
* Person unable to give informed consent
* Refusal to participate
* Participation in a study on a drug/medical device/care technique likely to affect cognitive functions

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
"Discrimination score" | Weeks: 2
  Comparison of the recognition score obtained in each of the experimental conditions to the recognition score obtained in the control condition The score = the Number of correct answer (0 to 15, the higher score means better outcome)

SECONDARY OUTCOMES:
"Geneva Music-Induced Affect Checklist" scale | Weeks: 2
  Analysis Geneva Music-Induced Affect Checklist scale results. It is composed of 4 sub-score dimensions such as valence, activation, tension (stress level) and pleasure (14 items scale 1: "not at all" to 5 "hugely, it's a qualitative scale)

CONTACTS AND LOCATIONS:
Overall Officials: Céline BORG, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (3):
- France (3):
  - CHU Grenoble, Grenoble
  - CHU de Saint-Etienne, Saint-Etienne
  - HCL, Villeurbanne

IPD SHARING:
Plan to Share IPD: No